CLINICAL TRIAL: NCT00913835
Title: Randomized Phase 2 Trial Investigating Liposomal Doxorubicin With or Without Anti-Platelet Derived Growth Factor Receptor-Alpha (PDGFRα) Monoclonal Antibody IMC-3G3 in Patients With Platinum-Refractory or Platinum-Resistant Advanced Ovarian Cancer
Brief Title: A Study of Liposomal Doxorubicin With or Without Olaratumab (IMC-3G3) in Platinum-Refractory or Resistant Advanced Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13899; 2009-009035-30 (EudraCT Number); CP15-0802 (Other: ImClone Systems); I5B-IE-JGDA (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Ovarian Neoplasms
Keywords: Liposomal Doxorubicin; IMC-3G3; 3G3; Platinum resistant; Platinum refractory; Ovary; Neoplasm; PDGFr
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — olaratumab; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olaratumab and Liposomal Doxorubicin (Experimental): Olaratumab and Liposomal Doxorubicin
  Interventions: Biological: Olaratumab; Drug: liposomal doxorubicin
- Liposomal Doxorubicin: Optional Olaratumab Monotherapy (Active Comparator): Liposomal Doxorubicin Monotherapy until disease progression. Upon disease progression the participant had the option to receive Olaratumab monotherapy.
  Interventions: Biological: Olaratumab; Drug: liposomal doxorubicin

INTERVENTIONS:
Biological: Olaratumab — 20 milligrams per kilogram (mg/kg) administered by intervenous (IV) infusion every 2 weeks (14 days). Treatment will continue until there is evidence of progressive disease (PD) or development of unacceptable toxicity
  Other Names: LY3012207; IMC-3G3
Drug: liposomal doxorubicin — 40 milligrams per square meter (mg/m²) administered according to the manufacture's instructions every 4 weeks (28 days). Treatment will continue until there is evidence of PD or development of unacceptable toxicity

SUMMARY:
The purpose of this study is to determine if participants with platinum-refractory or platinum-resistant advanced ovarian cancer have a better outcome when treated with Olaratumab (IMC-3G3) in combination with Liposomal Doxorubicin than when treated with Liposomal Doxorubicin alone.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the progression-free survival (PFS) in participants with platinum-refractory or platinum-resistant advanced ovarian cancer when treated with the monoclonal antibody Olaratumab in combination with liposomal doxorubicin versus liposomal doxorubicin alone.

ELIGIBILITY:
Inclusion Criteria:

* The participant has histologically or cytologically confirmed epithelial ovarian cancer, primary peritoneal carcinoma, fallopian tube cancer, or ovarian clear cell carcinoma
* The participant must have at least one of the following: a platinum-free interval of ≤12 months after the final dose of primary or subsequent platinum-based therapy (platinum-resistant), progression during primary or subsequent platinum-based therapy (platinum-refractory), or persistent radiographic disease after primary or subsequent platinum-based therapy (platinum-refractory)
* The participant has a pre-study echocardiogram or multigated acquisition (MUGA) scan with an actual left ventricular ejection fraction (LVEF) ≥50%, within 21 days prior to randomization
* The participant has at least one unidimensionally measurable target lesion [≥20 millimeters (mm) with conventional techniques, or ≥10 mm by spiral computed tomography (CT) or magnetic resonance imaging (MRI)], as defined by Response Evaluation Criteria in Solid Tumors, Version 1.0 (RECIST v1.0) guidelines. Tumors within a previously irradiated field will be designated as "nontarget" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* The participant has recovered to Grade ≤1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 3.0 (NCI-CTCAE v3.0) from the effects of recent surgery, radiotherapy, chemotherapy, hormonal therapy, or other targeted therapies for ovarian cancer, with the exception of alopecia or peripheral neuropathy (which must have resolved to ≤Grade 2). The exceptions for such effects are allowed lab values of ≤Grade 2 specified elsewhere in these inclusion criteria
* The participant has an Eastern Cooperative Oncology Group (ECOG) Performance Status score of ≤1 at study entry
* The participant has the ability to understand and the willingness to sign a written informed consent
* The participant has adequate hematological functions [absolute neutrophil count (ANC) ≥1200 cells/microliter (cells/μL), hemoglobin ≥9 grams/deciliter (g/dL), and platelets ≥100,000 cells/μL]
* The participant has adequate hepatic function as defined by total bilirubin ≤1.5 × the upper limit of normal (ULN), and aspartate transaminase (AST) and alanine transaminase (ALT) ≤3 × the ULN (or ≤5 × the ULN in the presence of known liver metastases)
* The participant has adequate renal function as defined by serum creatinine ≤1.5 × the institutional ULN. If creatinine is above the ULN, the participant's creatinine clearance is ≥60 milliliters/minute (mL/min)
* The participant has urinary protein ≤1+ on dipstick or routine urinalysis; if urine dipstick or routine analysis is ≥2+, a 24-hour urine for protein must demonstrate <1000 milligrams (mg) of protein to allow participation
* The participant must have adequate coagulation function as defined by International Normalized Ratio (INR) ≤1.5 and a partial thromboplastin time (PTT) ≤5seconds above ULN. Participants on anticoagulation must be on a stable dose of anticoagulant with a therapeutic INR and no active bleeding within 14 days prior to randomization, or on low molecular weight heparin AND have no pathological condition carrying a high risk of bleeding. Mild elevations of PTT of up to 1.5 × the ULN are acceptable, provided that, in the opinion of the investigator, they are related to ongoing use of coumarins [for example (e.g.), warfarin]
* The participant has a pre-study echocardiogram or MUGA scan with an actual LVEF ≥50%, within 21 days prior to randomization
* Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to randomization and for the duration of study participation

Exclusion Criteria:

* The participant has brain metastases or leptomeningeal disease
* The participant received more than one biologic and/or more than one hormonal therapy, administered either concomitantly with platinum-based therapy or separately
* The participant has a history of treatment with other agents targeting platelet derived growth factor (PDGF) or PDGF receptor (PDGFR)
* The participant has an increased level of cancer antigen-125 (CA-125) in the absence of concomitant clinical or radiographic progression
* The participant has received radiotherapy, chemotherapy, or biologic therapy directed at the malignant tumor within 3 weeks prior to randomization, or hormonal therapy directed at the malignant tumor within 1 week prior to randomization. Continuation of hormone replacement therapy is permitted
* The participant has a suspected impending bowel obstruction (including partial obstruction), based on clinical or radiographic data
* The participant has a history of allergic reactions attributed to compounds of chemical or biologic composition similar to that of IMC-3G3
* The participant has an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring parenteral antibiotics, symptomatic congestive heart failure,uncontrolled hypertension, clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* The participant has a history of another primary cancer, with the exception of: a) curatively resected nonmelanomatous skin cancer; b) curatively treated cervical carcinoma in-situ; or c) other primary solid tumor treated with curative intent and no known active disease present and no treatment administered during the last 3 years prior to randomization
* The participant is pregnant or lactating
* The participant has ongoing side effects ≥Grade 2 due to agents administered more than 28 days prior to randomization. The exceptions for such effects are allowed lab values and toxicities of ≤Grade 2, specified in the inclusion criteria
* The participant has unstable angina pectoris, angioplasty, cardiac stenting, or myocardial infarction 6 months prior to randomization
* The participant has participated in clinical trials of experimental agents within 28 days prior to randomization
* The participant has a history of uncontrolled hereditary or acquired bleeding or thrombotic disorders
* The participant has a serious or nonhealing active wound, ulcer, or bone fracture
* The participant has known human immunodeficiency virus positivity
* The participant had a major surgical procedure, an open biopsy, or significant traumatic injury within 28 days prior to randomization
* The participant has received an anthracycline for any indication in the past

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (6):
  - ImClone Investigational Site, Joliet, Illinois
  - ImClone Investigational Site, Indianapolis, Indiana
  - ImClone Investigational Site, Baltimore, Maryland
  - ImClone Investigational Site, Boston, Massachusetts
  - ImClone Investigational Site, Detroit, Michigan
  - ImClone Investigational Site, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] McGuire WP, Penson RT, Gore M, Herraez AC, Peterson P, Shahir A, Ilaria R Jr. Randomized phase II study of the PDGFRalpha antibody olaratumab plus liposomal doxorubicin versus liposomal doxorubicin alone in patients with platinum-refractory or platinum-resistant advanced ovarian cancer. BMC Cancer. 2018 Dec 27;18(1):1292. doi: 10.1186/s12885-018-5198-4. PMID 30591028

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants from liposomal doxorubicin (Lip Dox) treatment group who had progressive disease (PD) had the option to receive to Olaratumab (Olara) monotherapy. Participants who had evidence of PD, died in either period, or received optional Olaratumab monotherapy from liposomal doxorubicin monotherapy were considered to have completed the study.
Groups:
- Olaratumab + Liposomal Doxorubicin: 20 milligrams per kilogram (mg/kg) of Olaratumab was administered as an intravenous (IV) infusion every 2 weeks (14 days) until there was evidence of progressive disease (PD) or development of unacceptable toxicity.
  40 milligrams per square meter (mg/m²) of liposomal doxorubicin was administered according to the manufacturer's instructions every 4 weeks (28 days) until there was evidence of PD or development of unacceptable toxicity.
- Liposomal Doxorubicin: Optional Olaratumab Monotherapy: 40 mg/m² of liposomal doxorubicin was administered according to the manufacturer's instructions every 4 weeks (28 days). Treatment continued until there is evidence of PD or development of unacceptable toxicity up to 130 weeks.
  Upon disease progression the participant had the option to receive Olaratumab monotherapy.
Period: Olara+Lip Dox and Lip Dox Monotherapy
Arm/Group | Olaratumab + Liposomal Doxorubicin | Liposomal Doxorubicin: Optional Olaratumab Monotherapy
Started | 63 | 62
Received Any Study Drug | 62 | 61
Completed | 55 | 55
Not Completed | 8 | 7
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 4 | 3
Not completed — Off Study Treatment/Alive | 1 | 1
Period: Lip Dox: Olaratumab Monotherapy
Arm/Group | Olaratumab + Liposomal Doxorubicin | Liposomal Doxorubicin: Optional Olaratumab Monotherapy
Started | 0 | 28
Received at Least 1 Dose of Study Drug | 0 | 28
Completed | 0 | 25
Not Completed | 0 | 3
Not completed — Other | 0 | 3

BASELINE CHARACTERISTICS:
Population: Modified Intent to Treat (mITT) Population: All participants who were randomized and received any quantity of study drug.
Groups:
- Olaratumab and Liposomal Doxorubicin: 20 mg/kg of Olaratumab was administered as an IV infusion every 2 weeks (14 days) until there was evidence of PD or development of unacceptable toxicity up to 130 weeks.
  40 mg/m² of liposomal doxorubicin was administered according to the manufacturer's instructions every 4 weeks (28 days) until there was evidence of PD or development of unacceptable toxicity.
- Liposomal Doxorubicin: Optional Olaratumab Monotherapy: 40 mg/m² of liposomal doxorubicin was administered according to the manufacturer's instructions every 4 weeks (28 days). Treatment continued until there was evidence of PD or development of unacceptable toxicity up to 130 weeks.
  Upon disease progression the participant had the option to receive Olaratumab monotherapy.
- Total: Total of all reporting groups
Arm/Group | Olaratumab and Liposomal Doxorubicin | Liposomal Doxorubicin: Optional Olaratumab Monotherapy | Total
Number analyzed (Participants) | 62 | 61 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (10.07) | 59.8 (9.70) | 59.3 (9.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 61 | 123
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 6 | 7
  Not Hispanic or Latino | 61 | 54 | 115
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 3 | 4
  Black or African American | 5 | 1 | 6
  Native Hawaiian of Other Pacific Islander | 0 | 1 | 1
  White | 54 | 54 | 108
  Other | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 33 | 73
  United Kingdom | 17 | 14 | 31
  Spain | 5 | 14 | 19
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — ECOG PS classified participants according to their functional impairment.
  Participants
    0-Fully Active | 37 | 31 | 68
    1-ambulatory, able to do light/sedentary nature | 25 | 30 | 55
Stratification Factor [Count of Participants; unit: Participants] — Participants reaction to prior platinum treatment.
  Participants
    Platinum Refractory | 15 | 16 | 31
    Platinum Resistant | 47 | 45 | 92

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from the day of randomization to the first evidence of progression as defined by Response Evaluation Criteria in Solid Tumors version 1.0 (RECIST v1.0) criteria or death from any cause. Progressive Disease (PD) is a 20% increase over the smallest sum of target lesions or new lesions. Participants who died without a reported prior disease progression were considered to have progressed on the day of their death. Participants who did not progress and were subsequently lost to follow-up had their data censored at the day of last tumor assessment.
Time Frame: Randomization to Progressive Disease (PD) or Date of Death (Up to 35 Months)
Population: Modified Intent to Treat (mITT) Population: All randomized participants who received any amount of study drug. Participants censored: Olaratumab=13, Liposomal Doxorubicin=14.
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | Olaratumab and Liposomal Doxorubicin | Liposomal Doxorubicin: Optional Olaratumab Monotherapy
Number analyzed (Participants) | 62 | 61
weeks | 18.1 [8.7 to 27.0] | 17.3 [14.1 to 31.9]
Statistical Analysis 1: Comparison: Olaratumab and Liposomal Doxorubicin vs Liposomal Doxorubicin: Optional Olaratumab Monotherapy; Test type: Superiority or Other; p = 0.8049, Log Rank; Stratified by prior platinum treatment, platinum-refractory versus platinum-resistance reaction; Hazard Ratio (HR) = 1.054, 90% CI 2-sided [0.751 to 1.478]

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from first day of therapy to the date of death from any cause. Participants who were alive at the end of the follow-up period or were lost to follow-up, OS was censored on the last date the participant was known to be alive.
Time Frame: First Day of Therapy to Date of Death (Up to 35 Months)
Population: mITT Population: All randomized participants who received any amount of study drug. Participants censored: Olaratumab=21, Liposomal Doxorubicin=23.
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | Olaratumab and Liposomal Doxorubicin | Liposomal Doxorubicin: Optional Olaratumab Monotherapy
Number analyzed (Participants) | 62 | 61
weeks | 72.3 [52.4 to 86.7] | 70.6 [51.4 to 106.4]
Statistical Analysis 1: Comparison: Olaratumab and Liposomal Doxorubicin vs Liposomal Doxorubicin: Optional Olaratumab Monotherapy; Test type: Superiority or Other; p = 0.6346, Log Rank; Stratified by prior platinum treatment, platinum-refractory versus platinum-resistance reaction; Hazard Ratio (HR) = 1.115, 90% CI 2-sided [0.768 to 1.618]

3. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) [Objective Response Rate (ORR)]
Description: The percentage of participants with a best overall response of confirmed CR or PR defined using RECIST v1.0 criteria. CR is the disappearance of all target and non-target lesions and normalization of cancer antigen-125 (CA-125) levels. PR is defined as having a ≥30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. The percentage of participants with objective response was calculated as: (number of participants whose best overall response of CR or PR/number of participants treated) * 100.
Time Frame: Randomization to PD (Up to 35 Months)
Population: mITT Population: All randomized participants who received any amount of study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Olaratumab and Liposomal Doxorubicin | Liposomal Doxorubicin: Optional Olaratumab Monotherapy
Number analyzed (Participants) | 62 | 61
percentage of participants | 12.9 [6.6 to 22.1] | 16.4 [9.2 to 26.2]
Statistical Analysis 1: Comparison: Olaratumab and Liposomal Doxorubicin vs Liposomal Doxorubicin: Optional Olaratumab Monotherapy; Test type: Superiority or Other; p = 0.6190, Fisher Exact

4. Secondary Outcome: Median Duration of Response
Description: Duration of response is the interval from the date of initial CR or PR until the first date criteria for PD is met using RECIST v1.0 criteria, or initiation of other (or additional) antitumor therapy is first reported, or death due to any cause. CR is the disappearance of all target and non-target lesions and the normalization of tumor marker levels. PR is a ≥30% decrease in the sum of the LD of target lesions without new lesions and progression of non-target lesions. PD is a ≥20% increase in the sum of the LD of target lesions and/or unequivocal progression of existing non-target lesions and/or detection of 1 or more new lesions. Participants who did not relapse were censored on the day of their last tumor assessment.
Time Frame: Date of Initial CR or PR to PD (Up to 35 Months)
Population: All participants who achieved CR or PR. Participants censored: Olaratumab=2, Liposomal Doxorubicin=4.
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | Olaratumab and Liposomal Doxorubicin | Liposomal Doxorubicin: Optional Olaratumab Monotherapy
Number analyzed (Participants) | 8 | 10
weeks | 39.1 [26.1 to 56.1] | 16.9 [15.3 to NA] — Upper limit of confidence interval (CI) not estimable, did not reach the upper limit of CI.

5. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Who Died
Description: Reported are the number of participants with clinically significant events, defined as serious AEs (SAEs) and other non-serious AEs regardless of causality and those who died during treatment and during the 30-day post-dose follow-up. A summary of SAEs and other non-serious AEs regardless of causality is located in the Reported Adverse Events module of this report.
Time Frame: Baseline Up to End of Treatment and 30-day Post-dose Follow-up (Up to 35 Months)
Population: All randomized participants who received any amount of study drug.
Measure: Number; unit: participants
Groups:
- Liposomal Doxorubicin: 40 mg/m² of liposomal doxorubicin was administered according to the manufacturer's instructions every 4 weeks (28 days). Treatment continued until there was evidence of PD or development of unacceptable toxicity up to 130 weeks.
  Upon disease progression the participant had the option to receive Olaratumab monotherapy..
- Liposomal Doxorubicin: Optional Olaratumab Monotherapy: 40 mg/m² of liposomal doxorubicin was administered according to the manufacturer's instructions every 4 weeks (28 days). Treatment continued until there was evidence of PD or development of unacceptable toxicity followed by 20 mg/kg of Olaratumab administered as an IV infusion every 2 weeks (14 days) until there was evidence of PD or development of unacceptable toxicity up to 130 weeks.
Arm/Group | Olaratumab and Liposomal Doxorubicin | Liposomal Doxorubicin | Liposomal Doxorubicin: Optional Olaratumab Monotherapy
Number analyzed (Participants) | 62 | 61 | 28
participants
  SAEs | 27 | 23 | 14
  Other Non-SAEs | 62 | 60 | 27
  Deaths on treatment or within 30 days of last dose | 2 | 2 | 0

6. Secondary Outcome: Percentage of Participants With Anti-Olaratumab Antibodies
Description: Participants with Treatment Emergent (TE) anti-olaratumab antibodies were participants with a 4-fold increase (2 dilutions) increase over a positive baseline antibody titer or for a negative baseline titer, a participant with an increase from the baseline to a level of 1:20.
Time Frame: Baseline Up to 30-Day Postdose Follow-Up (Up To 35 Months)
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and evaluable post-baseline antibody data.
Measure: Number; unit: percentage of participants
Arm/Group | Olaratumab and Liposomal Doxorubicin | Liposomal Doxorubicin: Optional Olaratumab Monotherapy
Number analyzed (Participants) | 57 | 20
percentage of participants | 1.8 | 0

7. Secondary Outcome: PFS of Participants Who Received Olaratumab After Liposomal Doxorubicin Monotherapy (Descriptive Statistics for Safety and Efficacy for Participants Who Continue on Olaratumab Monotherapy Following Disease Progression on Liposomal Doxorubicin Monotherapy)
Description: PFS is defined as the time from start of Olaratumab monotherapy to the first evidence of progression as defined by RECIST v1.0 criteria or death from any cause. PD is a 20% increase over the smallest sum of target lesions or new lesions. Participants who died without a reported prior disease progression were considered to have progressed on the day of their death. Participants who did not progress and were subsequently lost to follow-up had their data censored at the day of last tumor assessment.
Time Frame: From Start of Olaratumab Monotherapy to PD or Date of Death (Up to 20 Weeks)
Population: Participants who received Olaratumab treatment after PD on liposomal doxorubicin monotherapy. Participants censored=4
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | Liposomal Doxorubicin: Optional Olaratumab Monotherapy
Number analyzed (Participants) | 28
weeks | 7.7 [7.1 to 10.4]

8. Secondary Outcome: Area Under the Curve (AUC) of Olaratumab
Time Frame: Prior to and 1 Hour (h) After Olaratumab Infusion in Cycles 1, 2, and 4 and 48 h or 72 h, 144 h, 240 h or 264 h and 336 h Post-dose in Cycles 1 and 4 (28-day Cycles)
Population: Zero participants were analyzed. An insufficient amount of samples were collected to derive this measure.
Arm/Group | Olaratumab and Liposomal Doxorubicin | Liposomal Doxorubicin | Liposomal Doxorubicin: Optional Olaratumab Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Maximum Concentration (Cmax) of Olaratumab
Time Frame: Prior to and 1 h after Olaratumab Infusion in Cycles 1, 2, and 4 and 48 h or 72 h, 144 h, 240 h or 264 h and 336 h Post-dose in Cycles 1 and 4 (28-day Cycles)
Population: Zero participants were analyzed. An insufficient amount of samples were collected to derive this measure.
Arm/Group | Olaratumab and Liposomal Doxorubicin | Liposomal Doxorubicin | Liposomal Doxorubicin: Optional Olaratumab Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Half-life (t1/2) of Olaratumab
Description: The time it takes to reduce the concentration of Olaratumab in the plasma by 50%.
Time Frame: as for outcome 9
Population: Zero participants were analyzed. An insufficient amount of samples were collected to derive this measure.
Arm/Group | Olaratumab and Liposomal Doxorubicin | Liposomal Doxorubicin | Liposomal Doxorubicin: Optional Olaratumab Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Clearance (CL) of Olaratumab
Description: CL is the volume of serum cleared of Olaratumab per unit of time after a single dose of Olaratumab
Time Frame: as for outcome 9
Population: Zero participants were analyzed. An insufficient amount of samples were collected to derive this measure.
Arm/Group | Olaratumab and Liposomal Doxorubicin | Liposomal Doxorubicin | Liposomal Doxorubicin: Optional Olaratumab Monotherapy
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Apparent Volume of Distribution (Vss) of Olaratumab
Description: Vss is an estimate of drug distribution independent of the elimination process and is proportional to the amount of drug in the body versus the drug plasma concentration at steady-state.
Time Frame: as for outcome 9
Population: Zero participants were analyzed. An insufficient amount of samples were collected to derive this measure.
Groups:
- Liposomal Doxorubicin: Optional Olaratumab Treatment: 40 mg/m² of liposomal doxorubicin was administered according to the manufacturer's instructions every 4 weeks (28 days). Treatment continued until there was evidence of PD or development Olaratumab administered as an IV infusion every 2 weeks (14 days) until there was evidence of PD or development of unacceptable toxicity up to 130 weeks.
Arm/Group | Olaratumab and Liposomal Doxorubicin | Liposomal Doxorubicin | Liposomal Doxorubicin: Optional Olaratumab Treatment
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: PFS for Participants Who Had Tissue Samples for Platelet Derived Growth Factor Receptor Alpha (PDGFRα) Expression Determined by Immunohistochemistry (IHC) (Association Between PDGFRα Tumor Expression and PFS)
Description: PFS is defined as the time from the day of randomization to the first evidence of progression as defined by RECIST v1.0 criteria or death from any cause. PD is a 20% increase over the smallest sum of target lesions or new lesions. Participants who died without a prior disease progression were considered to have progressed on the day of their death. Participants who did not progress and were subsequently lost to follow-up had their data censored at the day of last tumor assessment. PDGFRα protein expression at baseline in tumor cells is determined by IHC using H-Scores and a cut point of 0. Participants were considered to have a high relative expression when H-Score is >0 and a low relative expression when H-Score=0. H-Score was calculated by summing the percentage of cell staining at each intensity multiplied by the weighted intensity of staining. Staining intensity: 0 (no staining), 1+ (weak staining), 2+ (medium staining), 3+ (strongest staining). H-Scores could range from 0-300.
Time Frame: Randomization to PD or Date of Death (Up to 130 Weeks)
Population: All participants who had evaluable PDGFRα results.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Olaratumab and Liposomal Doxorubicin | Liposomal Doxorubicin
Number analyzed (Participants) | 54 | 47
weeks
  High Expression (n=41, 36) | 21.0 [8.7 to 34.1] | 17.3 [12.3 to 33.9]
  Low Expression (n=13,11) | 32.7 [7.6 to 41.3] | 24.0 [8.1 to 36.1]

ADVERSE EVENTS:
Arm/Group | Olaratumab and Liposomal Doxorubicin | Liposomal Doxorubicin | Liposomal Doxorubicin: Optional Olaratumab Monotherapy
Serious Adverse Events (participants affected / at risk) | 27/62 | 23/61 | 14/28
Other Adverse Events (participants affected / at risk) | 62/62 | 60/61 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaratumab and Liposomal Doxorubicin (N=62) | Liposomal Doxorubicin (N=61) | Liposomal Doxorubicin: Optional Olaratumab Monotherapy (N=28)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (4) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (4) | 0 (0) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 2 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3) | 2 (2)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0)
Extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 2 (2)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Bacillus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Incorrect drug administration duration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Bradyphrenia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaratumab and Liposomal Doxorubicin (N=62) | Liposomal Doxorubicin (N=61) | Liposomal Doxorubicin: Optional Olaratumab Monotherapy (N=28)
Anaemia (Blood and lymphatic system disorders) | 10 (21) | 13 (23) | 6 (8)
Leukopenia (Blood and lymphatic system disorders) | 6 (10) | 2 (2) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 4 (5) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 16 (67) | 8 (23) | 2 (3)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 14 (18) | 6 (8) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 15 (22) | 25 (35) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 4 (4) | 5 (6) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 10 (11) | 7 (8) | 2 (3)
Ascites (Gastrointestinal disorders) | 12 (17) | 6 (9) | 5 (6)
Constipation (Gastrointestinal disorders) | 32 (40) | 24 (33) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 19 (28) | 13 (16) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 8 (14) | 7 (7) | 7 (7)
Dysphagia (Gastrointestinal disorders) | 4 (5) | 3 (5) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 4 (5) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (7) | 6 (7) | 1 (1)
Nausea (Gastrointestinal disorders) | 35 (61) | 39 (61) | 13 (16)
Odynophagia (Gastrointestinal disorders) | 1 (2) | 4 (4) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 23 (40) | 16 (34) | 2 (2)
Vomiting (Gastrointestinal disorders) | 21 (41) | 18 (33) | 10 (12)
Asthenia (General disorders) | 8 (11) | 11 (21) | 4 (6)
Early satiety (General disorders) | 3 (3) | 4 (4) | 0 (0)
Fatigue (General disorders) | 33 (64) | 27 (50) | 5 (6)
Mucosal inflammation (General disorders) | 12 (19) | 15 (38) | 2 (3)
Oedema peripheral (General disorders) | 10 (13) | 12 (16) | 3 (3)
Pyrexia (General disorders) | 8 (15) | 7 (7) | 3 (3)
Candidiasis (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 2 (3) | 2 (3) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 4 (5) | 2 (2)
Urinary tract infection (Infections and infestations) | 15 (23) | 3 (5) | 3 (3)
Haemoglobin decreased (Investigations) | 7 (8) | 4 (4) | 2 (3)
Neutrophil count decreased (Investigations) | 3 (6) | 5 (5) | 0 (0)
Weight decreased (Investigations) | 9 (10) | 4 (4) | 1 (1)
White blood cell count decreased (Investigations) | 6 (27) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 15 (31) | 13 (19) | 10 (10)
Dehydration (Metabolism and nutrition disorders) | 7 (7) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (8) | 7 (8) | 4 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 (15) | 6 (8) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (13) | 7 (8) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (18) | 9 (12) | 5 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 (14) | 3 (3) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 9 (9) | 1 (2)
Dizziness (Nervous system disorders) | 10 (12) | 10 (13) | 1 (1)
Dysgeusia (Nervous system disorders) | 10 (12) | 3 (6) | 0 (0)
Headache (Nervous system disorders) | 12 (18) | 7 (8) | 6 (7)
Lethargy (Nervous system disorders) | 6 (10) | 4 (6) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 5 (6) | 2 (4) | 0 (0)
Paraesthesia (Nervous system disorders) | 3 (4) | 6 (7) | 0 (0)
Tremor (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 7 (7) | 6 (6) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (5) | 3 (3) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (3)
Pollakiuria (Renal and urinary disorders) | 4 (5) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 7 (10) | 2 (2) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 7 (7) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 10 (12) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (4) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (11) | 4 (4) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (11) | 9 (10) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 7 (11) | 7 (11) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (11) | 10 (11) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 7 (7) | 8 (10) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 21 (54) | 27 (60) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 24 (37) | 14 (34) | 4 (5)
Skin discolouration (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (4) | 6 (11) | 0 (0)
Flushing (Vascular disorders) | 4 (4) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 3 (3) | 1 (1)
Hypotension (Vascular disorders) | 4 (5) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.